CLINICAL TRIAL: NCT01531660
Title: Active Over 45: A Step-up Jogging Program in Inactive Female Hospital Staff Aged 45+: Feasability, Role of Motivation and Sustained Benefit
Brief Title: Active Over 45: A Step-up Jogging Program in Inactive Female Hospital Staff Aged 45+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Pierrette Baschung, MPH, MPH, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: active over 45
Record Dates: First submitted 2012-01-30; First posted 2012-02-13 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- training (Experimental): step up jogging program
  Interventions: Behavioral: step-up jogging program

INTERVENTIONS:
Behavioral: step-up jogging program

SUMMARY:
Background: Inactive individuals face motivational obstacles for becoming and staying physically active. Therefore, sustainable physical activity promotion programs tailored to reach inactive individuals are needed.

Purpose: to test the effect (long and short-term) and feasibility of a training program and to evaluate the association between the baseline motivation to become physical activity and the change in physical activity and performance.

Design: uncontrolled trail Setting/participants: inactive, female hospital staff aged 45 and older from the University Hospital Zurich Intervention: 3-month step-up jogging program Main outcome measures: physical performance and level of physical activity

ELIGIBILITY:
Inclusion criteria:

* female hospital stuff
* no regular physical activity
* older than 45 years

Exclusion criteria:

* osteoporotic fracture in the last three month
* significant musculoskeletal, cardiac or respiratory disorder

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-04; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
physical activity | 3 and 12 month
  Coopertest

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Daniel Uebelhart, MD, Principal Investigator — University Hospital Zurich, Division of Rheumatology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland